CLINICAL TRIAL: NCT02887170
Title: Recurrence of Suicide Attempt in Adolescents Lost to Contact Early by Clinicians : The 10-years REPEATERS Cohort of French Adolescents
Brief Title: The 10-years REPEATERS Cohort of French Adolescents
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Other Study IDs: u000420
Record Dates: First submitted 2016-08-24; First posted 2016-09-02 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Suicide Attempt
Keywords: Adolescent; Lost to contact; Recurrence; Long-term outcome
MeSH Terms: conditions — Suicide, Attempted; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Losing contact with adult suicide attempters in the year after the suicide attempt (SA) increases the risk of recurrence. The situation with adolescents is unknown. Investigators aimed to determine whether being lost to contact early (LCE) by clinicians is a risk factor of longterm SA recurrence among adolescents and the associated factors.

DETAILED DESCRIPTION:
Local clinical practice :

After an SA, adolescents receive treatment in the Children's Hospital or in the center of psychiatric consultation (few go to a private care clinic). All centers of psychiatric consultation belong to the same hospital center, which uses a unique medical record. According to the local clinical practice, patients and their parents systematically meet the child and adolescent psychiatric-department social worker at the time of the SA. The social worker informs the family that they will be called after 1 year to determine whether patients are safe or whether they need to resume care. For this call, the social worker uses the phone number listed in the medical record or finds the phone number in the national phone directory. If the social worker fails to contact the patient, the patient is considered LCE.

Patient follow-up :

Ten years after the index SA (every other year from 2004 to 2010), a self-reporting questionnaire will be sent to all adolescent suicide attempters and their parents, with a letter explaining the research. If the address of the patient is not available, the hospital records department will be contacted to collect these data for patients who will be re-hospitalized during the study period. When adolescent suicide attempters will be not contacted and when no information will be found in hospital records, the French Civil status Office will be called to determine whether patients were still alive. When no further information will be obtained, the adolescent will be considered lost to follow-up (LF) at the time of the last information from 1 to 10 years after the index SA.

Data collection :

At the time of the index SA, personal and family data will be collected from medical records for adolescents: personal characteristics (sex, age, history of SA [yes/no], psychiatric comorbidities of the SA [yes/no] according to the International Classification of Disease 10 (WHO, 1993), school difficulties [yes/no], and family characteristics (marital relationship of parents [separated or not], professional status of each parent [working or not], family history of SA [yes/no], and alcoholic dependence of parents [yes/no]). After the index SA, data on duration of hospitalization, psychiatric follow-up [yes/no], recurrence of SA in the year following the index SA (early SA recurrence [yes/no]), and LCE status [yes/no]) will be collected. Ten years after the index SA, a self-reporting questionnaire will be sent to the patient to assess SA recurrence.

ELIGIBILITY:
Inclusion Criteria:

* All adolescents who were hospitalized after an suicide attempt every other year from 1994 to 2000 in Nancy University Children's Hospital

Exclusion Criteria:

* The same patient being included twice

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all adolescents (ages 13e18 years old) who were hospitalized after an SA every other year from 1994 to 2000 in Nancy University Children's Hospital, were included without the same patient being included twice.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 1994-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
loss to contact after suicide attempt | one year

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne LIGIER, Principal Investigator — Nancy University Children's Hospital
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
open to partnership

REFERENCES:
- [Background] Ligier F, Guillemin F, Angot C, Bourion S, Kabuth B. Recurrence of suicide attempt in adolescents lost to contact early by clinicians: The 10-year REPEATERS cohort of French adolescents. J Adolesc. 2015 Aug;43:111-8. doi: 10.1016/j.adolescence.2015.05.011. Epub 2015 Jun 12. PMID 26073674